CLINICAL TRIAL: NCT01992692
Title: Remifentanil Requirement in Patients Receiving Surgical Treatment of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Jia-feng Wang, Dr., Changhai Hospital
Other Study IDs: Parkinson-remifentanil
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-06

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; remifentanil; deep brain stimulator; cardiovascular response
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PD group: Parkinsonian patients undergoing deep brain stimulator insertion and pulse generator placement
- non-PD group: Non-Parkinsonian patients undergoing intracranial surgery

SUMMARY:
Parkinson's disease (PD) is one the main neurodegenerative disease with an incidence of about 3% in patients older than 65 years. Anesthesia in PD patients has been focused by several studies for concerning the interactive reaction between anesthetics and anti-Parkinsonian medication or Parkinsonian symptoms. However, our previous experience showed that the patients undergoing pulse generator placement were more prone to be involved in delayed emergence in the recovery room, which had been not reported yet. We speculated that PD patients might be a special population with abnormal pharmacodynamic characters of anesthetics, though no related evidence could be found to support this hypothesis. Therefore, in this project we investigated whether remifentanl requirement to inhibit patients' response to trachea intubation and skin insertion in PD patients undergoing DBS and pulse generator placement was different from non-PD patients undergoing intracranial surgery for reasons other than PD.

ELIGIBILITY:
Inclusion Criteria:

* Adult Parkinsonian patients undergoing deep brain stimulator insertion and pulse generator placement
* Adult non-Parkinsonian patients undergoing intracranial surgery

Exclusion Criteria:

* ASA score higher than Class II
* predicted difficult airway
* alcohol or drug abuser
* informed consent was not provided

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinsonian patients undergoing deep brain stimulator insertion and pulse generator placement, as well as non-Parkinsonian patients undergoing intracranial surgery
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Concentrations required to inhibit response to trachea intubation and skin incision | Anesthesia induction to 5min after skin incision

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, Changhai Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Wang JF, Xu XP, Yu XY, Li JB, Wu X, Chen JC, Hu XW, Deng XM. Remifentanil Requirement for Inhibiting Responses to Tracheal Intubation and Skin Incision Is Reduced in Patients With Parkinson's Disease Undergoing Deep Brain Stimulator Implantation. J Neurosurg Anesthesiol. 2016 Oct;28(4):303-8. doi: 10.1097/ANA.0000000000000229. PMID 26368663